CLINICAL TRIAL: NCT06332274
Title: tislelizUMaB in canceR Patients With molEcuLar residuaL Disease
Acronym: UMBRELLA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: BeiGene (Industry); Veracyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-503316-33-00; 2023/3720 (Other: CSET number)
Record Dates: First submitted 2024-02-29; First posted 2024-03-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Lung Cancer; Colo-rectal Cancer; Pancreas Cancer; Soft Tissue Sarcoma
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Sarcoma | interventions — tislelizumab; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, randomized, placebo-controlled, multi-center, national, Phase 3 biology-driven trial designed to investigate the impact of systemic treatment with tislelizumab or placebo following detection of MRD minimum 3 months and maximum 4.5 months after completion of curative-intent therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A. MRD(+) - Tislelizumab treatment (Experimental): Systemic treatment with tislelizumab monotherapy at the recommended dose of 400 mg administered intravenously every 6 weeks for a maximum of 9 cycles and followed-up as per standard of care (clinical examination plus imaging every 3 months the first year and every 6 months the second year) in addition to ctDNA (circulating tumoral DNA) analysis at M6 and M12.
  Interventions: Drug: Tislelizumab; Other: Blood sampling
- Arm B. MRD(+) - placebo treatment (Placebo Comparator): Control arm for MRD (+) subjects who will be administered with placebo instead of tislelizumab
  Interventions: Other: Blood sampling; Drug: Placebo
- Arm C. MRD(-) - De-escalated follow-up (Experimental): De-escalated follow-up: clinical examination plus imaging every 6 months the first year and yearly the second year) with standard of care in addition to biobanking at M12 for subsequent ctDNA analyses.
  Interventions: Other: Blood sampling
- Arm D. MRD(-) - De-escalated follow-up (Other): Control arm for MRD (-) subjects , followed up as per standard of care (clinical examination plus imaging every 3 months the first year and every 6 months the second year) in addition to biobanking at M12 for subsequent ctDNA analyses.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Drug: Tislelizumab — Formulation : 100 mg of antibody in 10 mL of isotonic solution (25 mM citrate buffer, 15 mM L-histidine/histidine hydrochloride, 190 mM trehalose-dihydrate, and 0.02% polysorbate 20 at pH 6.5) in a single-use vial.
  Dose Regimen: Tislelizumab 400 mg every 6 weeks (Q6W) for a maximum of 9 cycles, on the first day of each cycle, in IV.
  Arms: Arm A. MRD(+) - Tislelizumab treatment
Other: Blood sampling — Blood sampling for analyses of MRD (Molecular Residual Disease)
Drug: Placebo — Pharmaceutical form : Solvent IV bags used for dilution of tislelizumab (for example: "CHLORURE DE SODIUM FRESENIUS 0,9 %, solution injectable") Dose Regimen: every 6 weeks (Q6W) for a maximum of 9 cycles, on the first day of each cycle, in IV.
  Arms: Arm B. MRD(+) - placebo treatment

SUMMARY:
Numerous studies have shown that even when imaging does not reveal the presence of cancer cells, traces of tumor DNA (i.e. originating from cancer cells) can be detected in the blood of certain patients: this is called molecular residual disease (MRD). When such traces are detected (we speak of MRD+ status), the risk of relapse is much higher than when there is no circulating tumor DNA (MRD - status). Given the success of immunotherapy in treating patients with metastatic disease in a variety of tumor types, there is enormous enthusiasm for expanding the use of immunotherapy to people with cancer at an early stage.

UMBRELLA is a biology-driven trial designed to study the impact of systemic treatment with tislelizumab monotherapy after detection of MRD+ status after completion of surgery and perioperative treatments in patients with cancer of a solid tumor. Residual disease (MRD) will be determined by optimized detection and precise monitoring of circulating tumor DNA, enabling early detection of recurrence and disease monitoring, including in patients without MRD [MRD(-)].

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Completion of surgical and peri-operative treatments as per international guidelines.
3. Subject must have completed standard curative-intent therapy (i.e: Surgery, Neoadjuvant and adjuvant therapy) for minimum 3 months and maximum 4.5 months prior to sending samples for MRD analyses.
4. Subject must not have standard treatment at least 3 weeks before blood sampling for ctDNA analyses.
5. Patients must not have blood transfusion at least 3 months before blood sampling for ctDNA analyses.
6. Histology: TNM stage II-III NSCLC, Stage II-III colorectal cancer, stage I-III pancreatic cancer, grade 3 limb or trunk wall soft-tissue sarcoma.
7. Subjects must have sufficient amount of archived primary tumor material for ctDNA and translational research analyses that will be conducted as defined in the protocol.
8. Subjects must have a valid (positive or negative) ctDNA test result prior to randomization.
9. Subjects must not have had prior immunotherapy (anti-PD-1 or anti-PD-L1).
10. No evidence of disease on imaging as per RECIST criteria 1.1.
11. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
12. Subjects must have adequate organ function as indicated by the following laboratory values (obtained within 7 days prior to randomization):

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, haemoglobin ≥90 g/L. Note: Patients must not have required growth factor support ≤ 14 days before sample collection.
    2. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x upper limit of normal (ULN).
    3. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
    4. Serum total bilirubin ≤ 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilbert's syndrome).
    5. Aspartate and alanine aminotransferase (AST and ALT) ≤ 3 x ULN.
    6. Creatinine clearance ≥60 mL/min for participants with creatinine levels above institutional normal (≥ULN). Creatinine clearance should be calculated per the Cockcroft-Gault formula (or local institutional standard method).
13. Subjects with a social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code).
14. Subjects should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
15. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the trial, and ≥ 120 days after the last dose of the trial drug and have a negative serum pregnancy test ≤ 7 days of the first dose of the trial drug. A barrier contraceptive method (e.g., condom) is also required. A woman is considered of childbearing potential following menarche and until becoming post-menopausal (≥ 12 months of non-therapy-induced amenorrhea) unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral oophorectomy and bilateral salpingectomy with surgery at least 1 month before the first dose of study drug or confirmed by follicle stimulating hormone (FSH) test >40 mIU/mL and estradiol <40 pg/mL (<140 pmol/L).
16. Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of the trial drug. A barrier contraceptive method (e.g., condom) is also required.

Exclusion Criteria:

1. Participation in another clinical trial with an investigational product during the last 3 to 4.5 months and while on study treatment
2. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in a clinical trial or which would jeopardize compliance with the protocol,
3. Pregnant or breastfeeding women
4. Subjects under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.
5. Patients with confirmed EGFR (Epidermal Growth Factor Receptor ) exon 19 deletions or exon 21 L858R substitutions are excluded from the study, due to the potential benefit from adjuvant osimertinib treatment, which represents a standard of care for these genetic profiles in non-small cell lung cancer (NSCLC).
6. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment
7. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate and thalidomide) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

   * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids as premedication for hypersensitivity reaction (e.g., CT scan premedication)) are eligible for the study after Principal investigator approval has been obtained
   * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
   * Patients who received intranasal, inhaled, topical or local steroid injections (e.g., intra articular injection)
8. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1.
9. Known intolerance the study drugs or any of their excipients
10. Patients with prior allogeneic stem cell or solid organ transplantation
11. Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study or within 5 months after the last dose of the study drugs (except anti-COVID-19 vaccines)
12. Active or history of autoimmune disease or immune deficiency, with the exception of history of treated autoimmune-related hypothyroidism and Type 1 diabetes mellitus on insulin regimen
13. History of idiopathic pulmonary fibrosis (including pneumonitis or interstitial lung disease), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis (history of radiation pneumonitis in the radiation field (fibrosis) is permitted).
14. Patients who underwent major surgery within 56 days prior to inclusion or until the surgical wound is fully healed
15. History of HIV infection
16. Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
17. Active tuberculosis.
18. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
19. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
20. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
21. Significant cardiovascular disease, such as:

    * History of myocardial infarction, acute coronary syndromes or coronary angioplasty/stenting/bypass grafting within the past 6 months,
    * Congestive Heart Failure (CHF) NYHA class III or IV or history of CHF NYHA class III or IV, unless an echocardiogram or multi-gated acquisition scan performed within 3 months day 1 reveals a left ventricular ejection fraction ≥ 55%
22. Uncontrolled hypertension defined by systolic pressure > 150 and/or diastolic pressure > 110 mmHg, with or without anti-hypertensive medication. Patients with initial blood pressure elevations are eligible if initiation or adjustment of anti-hypertensive medication lowers blood pressure to meet entry criteria
23. History of stroke or transient ischemic attack within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of tislelizumab compared to placebo as measured by DFS (Disease-free survival) | relapse/death assessed up to 60 months and at 12 months, 24 months, 48 months and 60 months.
  DFS for MRD (+) patients defined as the time from randomization to relapse or death, whichever occurs first. DFS rate will also be assessed at 12 months, 24 months, 48 months and 60 months.

SECONDARY OUTCOMES:
Estimation of DFS in subjects without MRD | relapse/death assessed up to 60 months
  DFS for MRD (-) patients defined as the time from randomization to relapse or death, whichever occurs first.
Estimation of overall survival (OS) | 12, 24, 48 and 60 months
Percentage of MRD (+) subject's completion of standard curative-intent therapy | 1 year after the end of enrollment
Time between detection of MRD and detection of relapse at imaging. | 1 year after the end of enrollment
  As documented per RECIST v1.1
Percentage of subjects with MRD assessment failure. | 1 year after the end of enrollment
Estimation of the time to become MRD (-) for MRD(+) patients | 1 year after the end of enrollment
  Time from baseline to detection of MRD (-) status in subjects who were MRD (+) at baseline
Evaluation of Health-Related Quality of Life (QLQ) by QLQ-C30 | Baseline and at months 6, 12, 18 and 24.
  Scores from EORTC QLQ-C30 (Quality of Life Questionnaire)
Evaluation of Health-Related Quality of Life (QLQ) by EQ-5D-5L | Baseline and at months 6, 12, 18 and 24.
  Scores from EuroQol EQ-5D-5L questionnaire
Cost effectiveness analysis: incremental cost | 1 year after the end of enrollment
Cost effectiveness analysis: QALY | 1 year after the end of enrollment
  Quality-Adjusted Life Year
Cost effectiveness analysis: ICER | 1 year after the end of enrollment
  Incremental Cost-Effectiveness Ratio (€/QALY).

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No